CLINICAL TRIAL: NCT01988766
Title: Risk of Central Venous Stenosis in Patients With Chronic Renal Failure After IJ Line Placement
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB12-1889
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Thrombosis
Keywords: Thrombosis; Central Venosis Catheter; Renal Disease; Vascular Access
MeSH Terms: conditions — Thrombosis; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Thrombosis: incidence of thrombosis in subjects who had PICC line placement
- No Thrombosis: no incidence of thrombosis in subjects who had PICC line placement

SUMMARY:
The purpose of this study is to compare the difference in thrombosis as a result of internal jugular (IJ) catheters versus peripherally inserted central catheter (PICC) lines. It is hypothesized that there will be a decreased rate of thrombosis in patients as a result of IJ catheters verses PICC lines.

DETAILED DESCRIPTION:
In a cohort of patients from Sept 1, 2010 until December 31, 2011 with chronic kidney disease (CKD) has shown that the incidence of IJ thrombosis after short term catheter access occurred in only 1/26 subjects or 4%. The current study is being done to compare this experience with the incidence of thrombosis from PICC lines. A secondary aim will be to determine if variables such as level of renal function, prior history of thrombosis or atherosclerosis contribute to the risk of thrombosis when PICC lines are placed. This data will provide the first comparison of the incidence of thrombotic complications from short term IJ catheter access versus PICC lines.

ELIGIBILITY:
Inclusion Criteria:

* subjects who had a PICC line placed at the University of Chicago between September 1, 2010 and December 31, 2011

Exclusion Criteria:

* subjects under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who had a PICC line placed at the University of Chicago by the procedure service between September 1, 2010 and December 31, 2011
Sampling Method: Non-Probability Sample
Enrollment: 1424 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Thrombosis | 15 months
  To calculate the incidence of deep venous thrombosis from PICC lines in patients

SECONDARY OUTCOMES:
Demographic Risk Factor Association with Risk of Thrombosis from PICC or IJ access | 15 months
  To evaluate if factors, known to be associated with thrombosis and atherosclerosis, are associated with the risk of thrombosis from PICC or IJ access. These factors include: renal failure, diabetes, hypertension, cancer, transplant, gender, age or the indication for the access, including antibiotics or chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Hammes, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States